CLINICAL TRIAL: NCT01979926
Title: Double-blind, A Multicenter, Randomized, Placebo-controlled, Parallel, Phase 2 Study to Comparative Evaluate the Efficacy of N02RS1 600mg/Day, 12,00mg/Day in Korean Patients With Acute and Chronic Bronchitis
Brief Title: Comparative Evaluate the Efficacy to Acute and Chronic Bronchitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PMK-N02RS1
Record Dates: First submitted 2013-10-31; First posted 2013-11-08 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Acute Exacerbation of Chronic Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- N02RS1 200mg (Experimental): Combination of Broussonetia spp and Lonicera spp
  Interventions: Drug: Combination of Broussonetia spp and Lonicera spp
- N02RS1 400mg (Experimental): Combination of Broussonetia spp and Lonicera spp
  Interventions: Drug: Combination of Broussonetia spp and Lonicera spp
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Drug: Combination of Broussonetia spp and Lonicera spp

INTERVENTIONS:
Drug: Combination of Broussonetia spp and Lonicera spp — 600 mg/ day or 1200 mg/ day for 7 days
  Other Names: N02RS1

SUMMARY:
The Purpose of A Multicenter, Randomized, Double-blind, Placebo-controlled to Evaluate the Efficacy, Safety and Pharmacokinetics of N02RS1 600mg and 1,200mg per day in Patients With acute and acute exacerbation of chronic bronchitis for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18, under 75 years of age
* Patients Acute and Chronic Bronchitis

Exclusion Criteria:

* Patients who have gotten a glucocorticoids treatment within 4 weeks.
* Patients who need treatments of antibiotic and acute bronchitis infection.
* Patients who have gotten teatments of antibiotic,bronchodilator,painkiller and secretagog within 7 days.
* Bronchial asthma patient.
* Patients who have an indication of bleeding.
* Patients who have a serious heart and renal disease or liver ailment or immunosuppressive response.
* Patients who have history of over 3 phage of Chronic obstructiv lung disease
* Bronchiectasis patients.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety | 12weeks
  1.Adverse Event: symptom, start day and time, end day and time, injection time, severity, progress, outcome, relation with investigational product.

SECONDARY OUTCOMES:
Efficacy | 12weeks
  1. Before and after physical examination
  2. Before and after bital Sign: blood pressure, pulse rate, temperature.
  3. Before and after Lanza Score at the duodenum and stomach
  4. Lab: hematologic examination, blood coagulation examination,urine examination
  5. Cumulative incidence rate of an endoscopic peptic ulcer.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne B An, Bs, Study Director — Korea Pharmaceutical Manufacturers Association
Locations (1):
- Seoul Nat'l University of Boramae Hospital, Seoul, Seoul, South Korea